CLINICAL TRIAL: NCT03030573
Title: Reconstruction of Postcholecystectomy Bile Duct Injury and Bile Duct Defects With the Round Ligament
Brief Title: Reconstruction of the Bile Duct With the Round Ligament
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beaujon Hospital (Other)
Responsible Party: Principal Investigator, Safi Dokmak, MD, Beaujon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beaujon Hospital
Record Dates: First submitted 2016-11-19; First posted 2017-01-25 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Bile Duct Obstruction, Extrahepatic
Keywords: Bile duct injury; Bile duct defect; Round ligament; Reconstruction
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device: Round ligament and the bile duct (Other): The investigators describe the safety and efficacy of the reconstruction of the bile duct with the Round ligament.
  Interventions: Procedure: Reconstruction of the bile duct with the round ligament

INTERVENTIONS:
Procedure: Reconstruction of the bile duct with the round ligament — In patients who had bile duct defect by injury or resection, the Round ligament will be used to reconstruct the defect. Surgical technique, the early and long term postoperative measures are detailed in the investigators protocol.

SUMMARY:
The investigators developed a new surgical technique in order to reconstruct the bile duct with the round ligament

DETAILED DESCRIPTION:
Classically, the bile duct defect after bile duct injury or resection is achieved by bilioenteric reconstruction. However bilioenteric anastomosis is associated with long term complications including intrahepatic bile ducts infection, specific complications related to the Roux en Y jejunal loop and eliminate the endoscopic access to intrahepatic bile ducts. The investigators had recently developed a new surgical technique to reconstruct the veins with the parietal peritoneum with excellent results. Accordingly the investigators decided to develop a new surgical technique in order to reconstruct the bile duct defects with the vascularized round ligament.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological or operative diagnosis of bile duct Injury or defect
2. Can underwent surgical procedure

Exclusion Criteria:

1) The absence of the round ligament

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Safety - absence of any severe complication or mortality related to the new procedure | at 1 year
  Safety is defined by the absence of any severe complication (necrosis or biliary fistula) or mortality related to the new procedure.

SECONDARY OUTCOMES:
Bile buct patency | at 3 year
  Secondary outcome include mainly the patency of the reconstructed bile duct.

CONTACTS AND LOCATIONS:
Overall Officials: Safi Dokmak, MD, Principal Investigator — HBP department, Beaujon hospital, Clichy, France
Locations (1):
- Departement HPB surgery, Beaujon Hospital, Clichy, Hauts de seine, France

IPD SHARING:
Plan to Share IPD: No